CLINICAL TRIAL: NCT06567613
Title: Validation of a Swiss German Language Test for Children
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University Hospital, Zürich (Other); Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00463; 5739 (Other: Inselspital Bern)
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Speech test — The hearing screening ensures normal hearing before enrollment. The speech reception threshold for swiss german mono- and bisyllable words is determined in an adaptive procedure.
  Other Names: Hearing screening

SUMMARY:
The aim of this study is to validate a Swiss German children's language test. Standard values for the speech intelligibility of Swiss German monosyllables and disyllables for children with normal hearing aged 4-6 years are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Native Swiss German speakers
* Hearing threshold better than 20dB HL at 0.5, 1, 2 and 4kHz
* Written informed consent by the parents

Exclusion Criteria:

* Hearing loss
* Cognitive impairment

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children without hearing loss
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Speech reception threshold for monosyllabic words | Single visit at baseline
  Speech Reception Threshold (SRT) measured in decibel sound pressure level (dB SPL), with lower scores indicating better hearing
Speech reception threshold for bisyllabic words | Single visit at baseline
  Speech Reception Threshold (SRT) measured in decibel sound pressure level (dB SPL), with lower scores indicating better hearing

SECONDARY OUTCOMES:
Speech reception threshold in noise for monosyllabic words | Single visit at baseline
  Speech Reception Threshold (SRT) measured in decibel signal-to-noise ratio (dB SNR) with lower scores indicating better hearing
Speech reception threshold in noise for bisyllabic words | Single visit at baseline
  Speech Reception Threshold (SRT) measured in decibel signal-to-noise ratio (dB SNR) with lower scores indicating better hearing

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schmid, Principal Investigator — Inselspital Bern, Berne University Hospital
Locations (4):
- Switzerland (4):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Luzern, Lucerne
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No
Data is only shared anonymously and aggregated